CLINICAL TRIAL: NCT06308289
Title: Combined Effects of Global Posture Re-education and Active Cycle of Breathing Technique on Cardiorespiratory Fitness, Posture and Quality of Life in Chronic Obstructive Pulmonary Disease
Brief Title: Combined Effects of Global Posture Re-education and Active Cycle of Breathing Technique in COPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/23/0361
Record Dates: First submitted 2024-03-04; First posted 2024-03-13 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-07

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: chronic obstructive Pulmonary disease; Posture; Work of breathing
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): GPRM and ACBT
  Interventions: Other: Global Posture Re-education; Other: Active Cycle of Breathing Technique
- Group B (Active Comparator): Standard Care for COPD (ACBT)
  Interventions: Other: Active Cycle of Breathing Technique

INTERVENTIONS:
Other: Global Posture Re-education — Focusing on postural correction and movement patterns
  Arms: Group A
Other: Active Cycle of Breathing Technique — Emphasizing breathing control, thoracic expansion, and mucus clearance techniques

SUMMARY:
The randomized controlled trial will involve 30 participants, with Group A receiving GPRM and ACBT, while Group B follows the conventional COPD model that includes ACBT only.Assessments of heart rate, physical fitness, and quality of life will contribute to a nuanced understanding of joint function, informing future COPD treatment paradigms.

DETAILED DESCRIPTION:
The focus of this study will be on addressing the critical challenge of treating chronic obstructive pulmonary disease (COPD), a globally prevalent and heterogeneous lung condition associated with substantial morbidity and mortality. With COPD anticipated to become the leading global cause of death, this research will investigate a novel intervention that combines global postural retraining (GPRM) and physical fitness, utilizing respiratory cycle technology (ACBT). This study assumes to enhance heart rate, posture, and overall quality of life in individuals with COPD. The randomized controlled trial will involve 30 participants, with Group A receiving GPRM and ACBT, while Group B follows the conventional COPD model that includes ACBT only. The study, utilizing nonprobability purposive sampling, will span six months to comprehensively evaluate cardiovascular, respiratory, and quality-of-life outcomes. Exclusion criteria ensure a representative sample, excluding individuals with severe diseases or recent surgeries. The significance of this investigation lies in its potential to revolutionize COPD treatment, offering a cost-effective approach that simultaneously enhances patient health. By targeting both biomechanical and respiratory aspects, the study aims to provide valuable insights into improving COPD treatment strategies globally, with a focus on the combined effects of global postural retraining and active breathing techniques. Assessments of heart rate, physical fitness, and quality of life will contribute to a nuanced understanding of joint function, informing future COPD treatment paradigms.

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged 40-75 years diagnosed with stable COPD (according to GOLD guidelines).
2. Patients of both genders
3. FEV1: FVC ranging from 68 - 69%.
4. Predicted FEV1 of less than 70%.
5. Willingness to participate

Exclusion Criteria:

1. Acute Exacerbation of COPD
2. Participants with severe comorbidities, such as unstable cardiovascular diseases (e.g., recent myocardial infarction, uncontrolled hypertension)
3. Participants diagnosed with respiratory conditions other than COPD (such as asthma, interstitial lung disease)
4. Individuals who have undergone major thoracic or abdominal surgery within the past three months
5. Individuals with severe mental health conditions (such as uncontrolled psychosis or severe depression)
6. Pregnant or lactating individuals.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2024-03-03 (Actual); Primary Completion 2024-06-05 (Actual); Study Completion 2024-06-15 (Actual)

PRIMARY OUTCOMES:
SF- 36 Questionnaire | 12 Weeks
  The 36-Item Short Form Survey (SF-36) is an outcome measure instrument that is often used, well-researched, self-reported measure of health. It stems from a study called the Medical Outcomes Study for the objective measure of the quality of life.
  It comprises 36 questions that cover eight domains of health:
  1. Limitations in physical activities because of health problems.
  2. Limitations in social activities because of physical or emotional problems
  3. Limitations in usual role activities because of physical health problems
  4. Bodily pain
  5. General mental health (psychological distress and well-being)
  6. Limitations in usual role activities because of emotional problems
  7. Vitality (energy and fatigue)
  8. General health perceptions Scores for the different domains are converted and pooled using a scoring key, for a total score indicating a range of low to high QOL
FEV1/FVC ratio | 12 Weeks
  The individual inhales maximally and then exhales forcefully into a spirometer, measuring lung volume and airflow. The procedure may be repeated multiple times to ensure accurate and consistent results.
6-minute walk test | 12 Weeks
  The Six-Minute Walk Test (6MWT) assesses exercise capacity. Participants are briefed and baseline vital signs are recorded.
  The 6 Minute Walk Test is a sub-maximal exercise test used to assess aerobic capacity and endurance. The distance covered over a time of 6 minutes is used as the outcome by which to compare changes in performance capacity.
Photogrammetry | 12 Weeks
  Photogrammetry is a research tool used in COPD studies to assess physical changes. It involves capturing and analyzing images of patients to measure anatomical features and body movement.
Forced expiratory volume (FEV1) | 12 Weeks
  The individual inhales maximally and then exhales forcefully into a spirometer, measuring lung volume and airflow. The procedure may be repeated multiple times to ensure accurate and consistent results.
Forced vital capacity (FVC) | 12 Weeks
  The individual inhales maximally and then exhales forcefully into a spirometer, measuring lung volume and airflow. The procedure may be repeated multiple times to ensure accurate and consistent results.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Faizan Hamid, MS-CPPT, Principal Investigator — Riphah International University
Locations (1):
- Social Security Hospital, Gujranwala, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No